CLINICAL TRIAL: NCT07265063
Title: Clinical and Radiographic Evaluation of Pulpotomy Using Calcium-Enriched Mixture Versus Pulpectomy Using Calcium Hydroxide/Iodoform Paste for the Treatment of Primary Molars With Irreversible Pulpitis: A Randomized Clinical Trial
Brief Title: Pulpotomy With CEM vs Pulpectomy With Ca(OH)2/Iodoform in Primary Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Hassab Elrasoul Abdelmagid Mohamed, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEMvsCHIP2025
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Carious Primary Molars
MeSH Terms: interventions — omega-Chloroacetophenone; Dental Cements; Metapex

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulpotomy Group (Experimental): Children in this group will undergo pulpotomy of second primary molars diagnosed with irreversible pulpitis using Calcium-Enriched Mixture (CEM) cement. The procedure includes coronal pulp removal, hemostasis, placement of CEM cement as a base over the pulp tissue, and final restoration with glass ionomer cement followed by stainless steel crown.
  Interventions: Procedure: Pulpotomy using Calcium-Enriched Mixture (CEM) Cement
- pulpectomy group (Experimental): Children in this group will undergo pulpectomy of second primary molars diagnosed with irreversible pulpitis using Calcium Hydroxide/Iodoform paste (Metapex). The procedure includes complete removal of the pulp tissue, canal instrumentation and irrigation, obturation with Metapex, and final restoration with glass ionomer cement followed by stainless steel crown.
  Interventions: Procedure: Pulpectomy using Calcium Hydroxide/Iodoform Paste (Metapex)

INTERVENTIONS:
Procedure: Pulpotomy using Calcium-Enriched Mixture (CEM) Cement — pulpotomy procedure using (CEM) Cement as pulp dressing material
  Arms: Pulpotomy Group
Procedure: Pulpectomy using Calcium Hydroxide/Iodoform Paste (Metapex) — pulpectomy procdure performed using Metapex paste as root canal filling material
  Arms: pulpectomy group

SUMMARY:
Will Calcium-Enriched Mixture (CEM) cement pulpotomy have less postoperative pain and more clinical and radiographic success compared to Calcium Hydroxide/Iodoform (Metapex) pulpectomy when managing second primary molars with irreversible pulpitis?

ELIGIBILITY:
Inclusion Criteria:

* Children:

Aged 6-8 years of both sexes. Cooperative and medically free. Diagnosed with irreversible pulpitis based on clinical and radiographic criteria.

Parents/legal guardians provide written informed consent. Parents able to attend follow-up visits.

Teeth:

Deep carious second primary molars with signs of irreversible pulpitis. No clinical signs of necrosis (abscess, fistula, mobility). No radiographic signs of necrosis (periapical lesion or resorption).

Exclusion Criteria:

* Children:

With systemic or mental disorders. Whose parents refuse to give consent. Uncooperative behavior.

Teeth:

Signs of pulpal necrosis (swelling, fistula, pathological mobility). Periapical or furcal radiolucency exceeding half the furcation-apical distance. Non-restorable teeth, root caries, internal/external resorption, or calcified canals.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Intensity | 1, 3, 6, 9, and 12 months post-treatment
  Pain intensity will be evaluated using the Visual Analog Scale (VAS) of faces, rated from 0 (no pain) to 5 (severe pain). Assessment will be performed at 1, 3, 6, 9, and 12 months after treatment. Clinical success will be considered when the patient reports no pain (score = 0).

SECONDARY OUTCOMES:
Evaluation of Clinical Success | 1, 3, 6, 9, and 12 months post-treatment
  Clinical success will be evaluated by the absence of pain, swelling, tenderness to percussion, sinus, fistula, and pathological mobility. Clinical assessment will be performed at 1, 3, 6, 9, and 12 months postoperatively.
Evaluation of Radiographic Success | 6 and 12 months post-treatment
  Radiographic success will be defined as the absence of widening of the periodontal ligament space, internal/external root resorption, or radiolucency in the furcation or periapical area. Radiographic failure will be recorded if any of these findings are observed.

IPD SHARING:
Plan to Share IPD: No